CLINICAL TRIAL: NCT02407366
Title: A Phase 2 Study of Icotinib With Concurrent Radiotherapy vs. Pemetrexed+ Carboplatin With Concurrent Radiotherapy in Unresectable Stage III Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor ( EGFR) Mutation
Brief Title: Icotinib With Concurrent Radiotherapy vs. Chemoradiotherapy in Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Guosheng Feng, Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGSLC-2015
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Inoperable stage III non-small cell lung cancer; EGFR mutation; Icotinib; Radiotherapy; Chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Icotinib with concurrent radiotherapy (Experimental): Icotinib (125 mg ,three times daily)with concurrent thoracic radiotherapy(TRT) (66 Gy/33 fractions), followed by maintenance icotinib (125 mg ,Three times daily) until disease progression or unacceptable toxicity.
  Interventions: Drug: Icotinib; Radiation: Thoracic radiotherapy(TRT)
- Chemoradiotherapy (Active Comparator): Pemetrexed(500mg/m2) + carboplatin (AUC，5) every 21 days for three cycles with concurrent thoracic radiotherapy(TRT) (66 Gy/33 fractions), followed by consolidation chemotherapy with two cycles of pemetrexed(500mg/m2) + carboplatin (AUC，5) every 21 days.Maintenance pemetrexed(500mg/m2) will be administered after consolidation chemotherapy until disease progression or unacceptable toxicity .
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Radiation: Thoracic radiotherapy(TRT)

INTERVENTIONS:
Drug: Icotinib — Icotinib (125 mg ,Three times daily)
  Other Names: BPI-2009; Conmana
  Arms: Icotinib with concurrent radiotherapy
Drug: Pemetrexed — Pemetrexed(500mg/m2)every 21 days
  Other Names: Alimta; LY231514; MTA; Multitargeted Antifolate; NSC-698037
  Arms: Chemoradiotherapy
Drug: Carboplatin — Carboplatin (AUC，5) every 21 days
  Other Names: Paraplatin
  Arms: Chemoradiotherapy
Radiation: Thoracic radiotherapy(TRT) — TRT (total dose 66Gy, 2Gy per time, once a day, five times a week, a total of 33 times)

SUMMARY:
The current standard of care for unresectable locally advanced non-small-cell lung cancer (NSCLC) is a combination of chemotherapy and thoracic radiotherapy (TRT). The standard regimens consist of platinum-based doublet chemotherapy.Icotinib(BPI-2009, Conmana) is the first self-developed small molecular drug in China for targeted therapy of lung cancer.Icotinib is a novel oral quinazoline compound that has proven survival benefit in Chinese patients with lung cancer,especially in EGFR mutation lung cancer. This randomised, multi-center, controlled trial is designed to assess the efficacy and safety of icotinib with concurrent radiotherapy versus pemetrexed + carboplatin with concurrent radiotherapy in inoperable stage III non-small cell lung cancer with EGFR mutation, the primary endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable stage IIIA / IIIB non-small cell lung cancer with EGFR 19/21 mutation.
2. No previous systemic anticancer therapy.
3. life expectancy more than three months.
4. ECOG Performance Status of 0 to 1.
5. Measurable lesion according to RECIST with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site.
6. Patients will be required to provide informed consent before enrollment.

Exclusion Criteria:

1. Intrapulmonary metastasis, atelectasis of an entire hemithorax,pleural dissemination, or contralateral hilar lymph node metastasis.
2. Prior chemotherapy for NSCLC, chest irradiation therapy, or therapy directed at the epidermal growth factor receptor pathway.
3. Severe heart disease, uncontrolled diabetes mellitus, or active infection.
4. Active concomitant malignancy, and pregnancy or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | One year
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival(OS) | two years
  Overall survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.
Adverse events | two years
  The number of patients who suffered adverse events, which is graded by NCI CTCAE version 4.0.
Objective response rate | two years
  Number of subjects with confirmed objective response according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Quality of life | two years
  Quality of life as measured by the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GuoSheng Feng, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; Yuan Liang, MD, Study Chair — Guangxi Department of Public Health; Lin Hui, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; HeMing Lu, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; ChangJie Huang, MD, Study Chair — Nanning Second People's Hospital; GuiSheng LI, MD, Study Chair — Liuzhou Workers' Hospital; HaiXin Huang, MD, Study Chair — Liuzhou Workers' Hospital; HaoLin Yan, MD, Study Chair — First People's Hospital of Yulin; Ping Liang, MD, Study Chair — Guangxi Ruikang Hospital; BingQiang Ni, MD, Study Chair — The People's hospital of LiuZhou; YanRong Hao, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; XianBin Yuan, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; Shan Gao, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; Xia Wu, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous; XiangLi Lai, MD, Study Chair — The People's hospital of Guangxi Zhuang Autonomous
Locations (1):
- The people's Hospital of the Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China